CLINICAL TRIAL: NCT02119741
Title: The Role of Hyaluronic Acid in Reconstruction of Interdental Papilla in The Esthetic Zone
Brief Title: Reconstruction of Interdental Papilla Using Hyaluronic Acid
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Perio-02-2014
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Defected Interdental Papilla
Keywords: Interdental papilla; hyaluronic acid; esthetic zone; black triangles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Affected Interdental Papillae Group: This is the only group in which the material will be used

SUMMARY:
Objective and background: The aim of this study is to evaluate the clinical outcome of using the hyaluronic acid gel in reconstructing inter-dental papillae at the aesthetic zones in a follow-up period of six months.

Materials and Methods: 30 interdental papilla deficiencies which would meet the the inclusion criteria will be evaluated. After applying local anesthesia, 0.2 ml hyaluronic acid gel will be injected at the affected areas. This procedure will be repeated 3 times for the evaluated areas. Photographs will be taken before injection this material, and at 3 and 6 months following the intervention.

DETAILED DESCRIPTION:
The presence or absence of the interproximal papilla is essential concern to periodontists, restorative dentists, and to the patients. The loss of papilla can cause cosmetic deformities (black triangles), phonetic problems, and food debris accumulation. Often the loss of papilla is a consequence of periodontal disease because of gingival inflammation, attachment loss and interproximal bone height resorption.

Several reasons also lead to absence of interdental papillae including:

1) Plaque associated lesions, 2) Traumatic oral hygiene procedures, 3) Abnormal tooth shape, 4) Improper contours of the restoration, 5) Spacing between teeth, 6) Loss of teeth.

ELIGIBILITY:
Inclusion Criteria:

The patient should be:

* 20-35 years old.
* Healthy with no systemic diseases.
* Non-smoker and non-alcoholic.
* with good oral hygiene.
* with healthy periodontal tissues.
* suffering from one defected interdental papilla at least.

Defected interdental papilla criteria:

* Class 2 according to Jemt Classification (Jemt 1997).
* The contact points between the teeth should be present.
* There are no restorations or caries in the adjacent teeth.
* The distance between the contact point and the interdental bone crest ≤ 6mm assessed radiographically.

Exclusion Criteria:

* History of allergic reaction to Hyaluronic acid
* Parafunctional habits.
* Traumatic occlusion.
* The patient under orthodontic treatment.
* Pregnant and lactating women.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the database of Periodontics Department at University of Damascus. A random sample of 30 patients will be included in this evaluation study from those who have been identified with defected interdental papillae.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of change in papillary height (PCPH) from baseline measurement | T0: baseline assessment, T1: immed. following injection, T2: after 3 weeks, T3: immed. following 2nd injection if required, T4: after 6 weeks from T1, T5: immed. following 3rd injection if needed, T6: after 3 months, T7: after 6 months postoperatively.
  The treated sites will be examined, defect measurements will be recorded, and photographs will be taken at a standard (1:1) magnification.
  The measurement of the distance from the tip of the interdental papilla to the base of the contact area for each study lesion separately using specific software.

SECONDARY OUTCOMES:
Change in the Interdental Papilla Index Score (CPIS) from baseline measurement | T0: baseline assessment, T1: immed. following injection, T2: after 3 weeks, T3: immed. following 2nd injection if required, T4: after 6 weeks from T1, T5: immed. following 3rd injection if needed, T6: after 3 months, T7: after 6 months postoperatively.
  The treated sites will be examined clinically, using a periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Ata Dalal, DDS, Principal Investigator — MSc student, Department of Periodontology, University of Damascus Dental School; Suleiman Dayoub, DDS MSc PhD, Study Director — Associate Professor of Periodontics, Department of Periodontics, University of Damascus Dental School, Damascus
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Agudio G, Pini Prato GP, Nevins M, Cortellini P, Ono Y. Esthetic modifications in periodontal therapy. Int J Periodontics Restorative Dent. 1989;9(4):288-99. No abstract available. PMID 2640208
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Angelopoulos AP, Goaz PW. Incidence of diphenylhydantoin gingival hyperplasia. Oral Surg Oral Med Oral Pathol. 1972 Dec;34(6):898-906. doi: 10.1016/0030-4220(72)90228-9. No abstract available. PMID 4509004
- [Background] Becker W, Gabitov I, Stepanov M, Kois J, Smidt A, Becker BE. Minimally invasive treatment for papillae deficiencies in the esthetic zone: a pilot study. Clin Implant Dent Relat Res. 2010 Mar;12(1):1-8. doi: 10.1111/j.1708-8208.2009.00247.x. Epub 2009 Oct 16. PMID 19843105
- [Background] Biesman B. Soft tissue augmentation using Restylane. Facial Plast Surg. 2004 May;20(2):171-7; discussion 178-9. doi: 10.1055/s-2004-861760. PMID 15643586
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid fillers: Restylane and Perlane. Facial Plast Surg Clin North Am. 2007 Feb;15(1):63-76, vii. doi: 10.1016/j.fsc.2006.11.002. PMID 17317557
- [Background] Jemt T. Regeneration of gingival papillae after single-implant treatment. Int J Periodontics Restorative Dent. 1997 Aug;17(4):326-33. PMID 9497723